CLINICAL TRIAL: NCT05564104
Title: A Study Investigating the Pharmacokinetic Properties of Cagrilintide in Participants With Various Degrees of Hepatic Impairment and Assessing the Absolute Bioavailability of Subcutaneous Cagrilintide in Healthy Volunteers
Brief Title: A Research Study Looking at How a Single Dose of the Medicine Cagrilintide Works in Participants With Reduced Liver Function and in Healthy Participants With Normal Liver Function and How Cagrilintide is Absorbed and Used by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9838-4692; U1111-1271-9259 (Other: World Health Organization (WHO)); 2022-000138-41 (EudraCT Number)
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hepatic Impairment; Healthy Volunteers
MeSH Terms: interventions — cagrilintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Participants with normal hepatic function (Experimental): Participants with normal hepatic function will receive a single subcutaneous (s.c.) dose of 0.9 milligrams (mg) of cagrilintide on Day 1.
  Interventions: Drug: Cagrilintide
- Part A: Participants with mild hepatic impairment (Experimental): Participants with mild hepatic impairment (Child Pugh Grade A) will receive a single subcutaneous (s.c.) dose of 0.9 milligrams (mg) of cagrilintide on Day 1.
  Interventions: Drug: Cagrilintide
- Part A: Participants with moderate hepatic impairment (Experimental): Participants with moderate hepatic impairment (Child-Pugh Grade B) will receive a single subcutaneous (s.c.) dose of 0.9 milligrams (mg) of cagrilintide on Day 1.
  Interventions: Drug: Cagrilintide
- Part A: Participants with severe hepatic impairment (Experimental): Participants with severe hepatic impairment (Child-Pugh Grade C) will receive a single subcutaneous (s.c.) dose of 0.9 milligrams (mg) of cagrilintide on Day 1.
  Interventions: Drug: Cagrilintide
- Part B: Sequence 1 (Experimental): Healthy participants will receive a single dose of cagrilintide Dose 1 intravenously (i.v) at the first dosing visit (Day 1), followed by a single dose of cagrilintide Dose 2 s.c. at the second dosing visit (Day 53).
  Interventions: Drug: Cagrilintide
- Part B: Sequence 2 (Experimental): Healthy participants will receive a single dose of cagrilintide Dose 2 s.c. at the first dosing visit (Day 1), followed by a single dose of cagrilintide Dose 1 i.v at the second dosing visit (Day 53).
  Interventions: Drug: Cagrilintide

INTERVENTIONS:
Drug: Cagrilintide — Cagrilintide will be administered subcutaneously in the abdomen in the form of a solution for injection as well as intravenously in the form of solution for injection.
  Other Names: NNC0174-0833

SUMMARY:
The study is divided into two parts - Part A and Part B. Cagrilintide in combination with semaglutide, is under development for weight management. In the development of cagrilintide, it is important to see if liver function influences how the body absorbs, breaks down, and eliminates cagrilintide (Part A) and also how the medicine is absorbed and used by the body in healthy participants (Part B). In Part A, this will be tested by comparing the blood levels of cagrilintide in participants with reduced liver function to those of participants with normal liver function and in Part B, it will be tested how this medicine is absorbed and used by comparing blood levels between participants who take the study medicine in different ways. Cagrilintide is a long-acting study medicine that resembles one of the body's own hormones called amylin that is involved in regulation of food intake and body weight. It is the hope that cagrilintide can help participants with weight management. Both the participant and the study doctor will know what treatment is being provided to the participant. In Part A, all participants will receive a single dose of 0.9 milligrams (mg)cagrilintide. The study medicine will be given in the form of an injection in a skinfold of the belly (subcutaneous) and in Part B, all participants will receive the same study medicine, taken in two different ways. Participants will get cagrilintide injected into your vein (intravenously) and injected under the skin (subcutaneously). Which treatment participants get first is decided by chance. The study will last up to 10 weeks in Part A and 91 days in Part B. If participants are eligible for this study, they will come to the clinic a total of 7 times and stay in the clinic for 7 days (6 nights) in Part A and in Part B, participants will stay in the clinic twice for a total of 12 days (10 nights). Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period. Women who are able to become pregnant must use highly effective contraception and will be counselled on the use of contraception.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Part A: Aged 18-80 years (both inclusive) at the time of signing informed consent.
* Part B: Aged 18-60 years (both inclusive) at the time of signing informed consent.
* Part A: Body mass index (BMI) between 18.5-39.9 kilograms per meter square (kg/m^2) (both inclusive).
* Part B: BMI between 25-30 kg/m2 (both inclusive).
* Specific inclusion criterion only for Part A participants with hepatic impairment: Participants with stable hepatic impairment classified as Child-Pugh grade A, B or C as assessed by the investigator. Stable hepatic impairment is defined as no clinically significant change in disease status, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Part A: AUC 0-infinity (∞), single dose (SD), cagri: The area under the cagrilintide plasma concentration-time curve fromtime 0 to infinity after a single dose | From 00 hours (pre-dose), 04, 08, 12, 18, 24, 30, 36, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 840 hours (post dose)
  Measured in nanomoles * hours per liter (nmol*h/L)

SECONDARY OUTCOMES:
Part A: Cmax,SD,cagri: Maximum observed plasma cagrilintide concentration after a single dose | From 00 hours (pre-dose), 04, 08, 12, 18, 24, 30, 36, 48, 54, 60, 72, 84, 96 to 120 hours (post dose)
  Measured in nanomoles per liter (nmol/L).
Part A: Tmax,SD,cagri: Time to maximum observed plasma cagrilintide concentration after a single dose | From 00 hours (pre-dose), 04, 08, 12, 18, 24, 30, 36, 48, 54, 60, 72, 84, 96 to 120 hours (post dose)
  Measured in hours (h).
Part A: T½ SD,cagri:Terminal half-life for cagrilintide after a single dose | From 00 hours (pre-dose), 04, 08, 12, 18, 24, 30, 36, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 840 hours (post dose)
  Measured in hours (h).
Part A: CL/F SD,cagri:Apparent clearance of cagrilintide after a single dose | From 00 hours (pre-dose), 04, 08, 12, 18, 24, 30, 36, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 840 hours (post dose)
  Measured in liters per hour (L/h).
Part B: AUC0-∞,SD,cagri: The area under the cagrilintide plasma concentration-time curve from time 0 to infinity after a single dose | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 912 hours (post dose)
  Measured in nmol*h/L
Part B: AUC0-last,SD,cagri: The area under the cagrilintide plasma concentration-time curve from time 0 to last quantifiable observation | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 912 hours (post dose)
  Measured in nmol*h/L
Part B: Cmax,SD,cagri: Maximum observed plasma cagrilintide concentration after a single dose | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96 to 120 hours (post dose)
  Measured in nmol/L
Part B: tmax,SD,cagri: Time to maximum observed plasma cagrilintide concentration after a single dose | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96 to 120 hours (post dose)
  Measured in hours (h)
Part B: t½ SD,cagri: Terminal half-life for cagrilintide after a single dose | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 912 hours (post dose)
  Measured in hours (h).
Part B: CL/F SD,cagri: Apparent clearance of cagrilintide after a single s.c. dose | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 912 hours (post dose)
  Measured in L/h.
Part B: CL SD,cagri: Apparent clearance of cagrilintide after a single i.v. dose | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 912 hours (post dose)
  Measured in L/h.
Part B: V z/F,cagri: Volume of distribution of cagrilintide after a single s.c. dose | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 912 hours (post dose)
  Measured in liters (L).
Part B: V z,cagri: Volume of distribution of cagrilintide after a single i.v. dose | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 912 hours (post dose)
  Measured in liters (L).
Part B: MRT SD,cagri: Mean residence time of cagrilintide | From 00 hours (pre-dose), 05 mins, 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 30 mins, 02, 02 hours 30 mins, 03, 04, 05, 06, 08, 10, 12, 16, 18, 20, 24, 30, 36, 42, 48, 54, 60, 72, 84, 96, 120, 168, 336, 504, 672 to 912 hours (post dose)
  Measured in hours (h).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (4):
- Pharmaceutical Research Associates CZ, s.r.o., Prague, Czechia
- APEX Research, München, Germany
- Slovakia (2):
  - Summit Clinical Research s.r.o., Bratislava
  - Summit Clinical Research s.r.o., Malacky

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com